CLINICAL TRIAL: NCT03800758
Title: A Randomized Controlled Trial Testing Expressive Helping for Stem Cell Transplant Patients
Brief Title: Expressive Helping for Stem Cell Transplant Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Lombardi Comprehensive Cancer Center (Other); Hackensack Meridian Health (Other)
Responsible Party: Principal Investigator, Christine Rini, PhD, Director, Cancer Survivorship Institute, Robert H. Lurie Comprehensive Cancer Center, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: PRO2018-0953; R01CA223963 (NIH); 2018-1306 (Other: Georgetown University)
Record Dates: First submitted 2019-01-08; First posted 2019-01-11 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-05

CONDITIONS: Stem Cell Transplantation; Hematologic Malignancy
MeSH Terms: conditions — Hematologic Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Expressive Helping writing (Experimental): Writing sessions 1-3: Participants complete one 20-minute expressive writing session at three time points: 1) after hospitalization but prior to transplant infusion, (2) approximately 3 days after hospital discharge, and (3) approximately 2 weeks after completion of writing session 2.
  Writing session 4: One 20-40 minute peer support writing session about 1 week after completion of writing session 3.
  Interventions: Behavioral: Expressive Helping
- Factual Writing (Active Comparator): Writing sessions 1-3: Participants complete one 20-minute factual session at three time points: 1) after hospitalization but prior to transplant infusion, (2) approximately 3 days after hospital discharge, and (3) approximately 2 weeks after completion of writing session 2.
  Writing session 4: One 20-40 minute factual writing session about 1 week after completion of writing session 3.
  Interventions: Behavioral: Factual Writing

INTERVENTIONS:
Behavioral: Expressive Helping — Expressive Helping (EH) is completed in 4 brief structured writing sessions during and immediately after transplant, with instructions focused on having participants write about their transplant experience using previously-tested EH instructions, adapted for this population.
  Arms: Expressive Helping writing
Behavioral: Factual Writing — Factual Writing has been used with cancer patients and in the investigators' prior EH trial. It is completed in 4 brief structured writing sessions during and immediately after transplant, with instructions focused on having participants write about their transplant experience using standard Factual Writing instructions.
  Arms: Factual Writing

SUMMARY:
The Writing for Insight, Strength, and Ease (WISE) Study is a multisite Randomized Controlled Trial (RCT) testing the efficacy of the Expressive Helping (EH) intervention among adults receiving hematopoietic stem cell transplantation.

DETAILED DESCRIPTION:
Use of stem cell transplant (mostly for hematologic cancers) is expected to increase 5-fold by 2030, when the number of survivors will reach 500,000. This highly toxic treatment causes a range of acute physical and psychological symptoms, which then persist for years for up to 45% of patients. To address gaps in existing symptom-focused behavioral interventions that can be added to standard patient care, the investigators developed Expressive Helping (EH), a low-cost, low-burden intervention that targets a range of physical and psychological symptoms in a broad group of transplant recipients. EH is completed in 4 brief structured writing sessions during and immediately after transplant, with instructions focused on having participants write about their transplant experience. Based on promising preliminary data, the investigators propose to determine whether EH can be used during and immediately after transplant to reduce common acute physical and psychological symptoms and prevent development of persistent physical and psychological symptoms. Assessments of physical symptoms and psychological symptoms will occur at baseline (prior to randomization), "nadir" (Day 7 post-transplant), "engraftment" (Day 14 post-transplant), 1 week post-intervention, 3-months post-intervention (primary endpoint, early post-transplant), 6-months post-intervention, and 12-months post-intervention (primary endpoint, later post-transplant). The investigators will also assess a select set of potential mediators and moderators of intervention effects. Participants will be adult cancer patients scheduled for allogeneic or autologous stem cell transplant at the study sites. After screening and consent, eligible patients will be enrolled in a parallel-group, 1:1 randomized controlled trial. Randomization will be stratified by study site (JTCC, Lombardi Comprehensive Cancer Center, LCCC, or Robert H. Lurie Comprehensive Cancer Center, RHLCCC); sex (linked with patient outcomes), age (18-59, ≥ 60), and transplant type (autologous, allogeneic). Staff performing assessments will be blind to study assignment. Participants cannot be blinded, but hypotheses will not be revealed to them until trial completion. They will be asked not to reveal their assignment to staff.

ELIGIBILITY:
Inclusion Criteria:

* Cancer patients
* Age ≥ 18
* English proficient
* Scheduled for allogeneic or autologous transplant at JTCC, LCCC, or RHLCC.

Exclusion Criteria:

* Current participation in a behavioral intervention targeting symptoms or quality of life
* Cognitive or psychiatric impairment precluding ability to complete informed consent or study procedures
* Literacy limitations precluding completion of a writing study
* Undergoing a tandem transplant where participant is now completing the first of two or more planned transplants

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 405 (Actual)
Dates: Start 2019-03-06 (Actual); Primary Completion 2023-04-24 (Actual); Study Completion 2023-04-24 (Actual)

PRIMARY OUTCOMES:
Symptom severity: Changes in symptom burden | Baseline to 3-months post intervention
  MD Anderson Symptom Inventory-Bone Marrow Transplant (MDASI-BMT), which measures both the severity of and interference caused by 13 symptoms, plus 5 transplant-specific symptoms. Symptom severity is rated on a 0-10 scale (0="not present" to 10="As bad as you can imagine") to indicate the severity of symptoms in the past 24 hours. The mean of items are calculated to yield a symptom severity score in which higher scores indicate higher severity.
Symptom severity: Changes in symptom burden | Baseline to 12-months post-intervention
  MD Anderson Symptom Inventory-Bone Marrow Transplant (MDASI-BMT), which measures both the severity of and interference caused by 13 symptoms, plus 5 transplant-specific symptoms. Symptom severity is rated on a 0-10 scale (0="not present" to 10="As bad as you can imagine") to indicate the severity of symptoms in the past 24 hours. The mean of items are calculated to yield a symptom severity score in which higher scores indicate higher severity.

SECONDARY OUTCOMES:
Symptom severity: Changes in symptom burden | Baseline to Day 7 post-transplant
  MD Anderson Symptom Inventory-Bone Marrow Transplant (MDASI-BMT), which measures both the severity of and interference caused by 13 symptoms, plus 5 transplant-specific symptoms. Symptom severity is rated on a 0-10 scale (0="not present" to 10="As bad as you can imagine") to indicate the severity of symptoms in the past 24 hours. The mean of items are calculated to yield a symptom severity score in which higher scores indicate higher severity.
Symptom severity: Changes in symptom burden | Baseline to Day 14 post-transplant
  MD Anderson Symptom Inventory-Bone Marrow Transplant (MDASI-BMT), which measures both the severity of and interference caused by 13 symptoms, plus 5 transplant-specific symptoms. Symptom severity is rated on a 0-10 scale (0="not present" to 10="As bad as you can imagine") to indicate the severity of symptoms in the past 24 hours. The mean of items are calculated to yield a symptom severity score in which higher scores indicate higher severity.
Symptom severity: Changes in symptom burden | Baseline to 1-week post-intervention
  MD Anderson Symptom Inventory-Bone Marrow Transplant (MDASI-BMT), which measures both the severity of and interference caused by 13 symptoms, plus 5 transplant-specific symptoms. Symptom severity is rated on a 0-10 scale (0="not present" to 10="As bad as you can imagine") to indicate the severity of symptoms in the past 24 hours. The mean of items are calculated to yield a symptom severity score in which higher scores indicate higher severity.
Symptom severity: Changes in symptom burden | Baseline to 6-months post-intervention
  MD Anderson Symptom Inventory-Bone Marrow Transplant (MDASI-BMT), which measures both the severity of and interference caused by 13 symptoms, plus 5 transplant-specific symptoms. Symptom severity is rated on a 0-10 scale (0="not present" to 10="As bad as you can imagine") to indicate the severity of symptoms in the past 24 hours. The mean of items are calculated to yield a symptom severity score in which higher scores indicate higher severity.
Depressive symptoms: Changes in depressive symptoms | Baseline to Day 7 post-transplant
  Center for Epidemiologic Studies Depression Scale (CES-D), is a 20-item measure that asks respondents to rate how often over the past week they experienced symptoms associated with depression on a scale from 0 to 3 (0 = "Rarely or None of the Time," 1 = "Some or Little of the Time," 2 = "Moderately or Much of the time," 3 = "Most or Almost All the Time"). Scores are summed and range from 0 to 60, with high scores indicating greater depressive symptoms.
Depressive symptoms: Changes in depressive symptoms | Baseline to Day 14 post-transplant
  Center for Epidemiologic Studies Depression Scale (CES-D), is a 20-item measure that asks respondents to rate how often over the past week they experienced symptoms associated with depression on a scale from 0 to 3 (0 = "Rarely or None of the Time," 1 = "Some or Little of the Time," 2 = "Moderately or Much of the time," 3 = "Most or Almost All the Time"). Scores are summed and range from 0 to 60, with high scores indicating greater depressive symptoms.
Depressive symptoms: Changes in depressive symptoms | Baseline to 1-week post-intervention
  Center for Epidemiologic Studies Depression Scale (CES-D), is a 20-item measure that asks respondents to rate how often over the past week they experienced symptoms associated with depression on a scale from 0 to 3 (0 = "Rarely or None of the Time," 1 = "Some or Little of the Time," 2 = "Moderately or Much of the time," 3 = "Most or Almost All the Time"). Scores are summed and range from 0 to 60, with high scores indicating greater depressive symptoms.
Depressive symptoms: Changes in depressive symptoms | Baseline to 3-months post-intervention
  Center for Epidemiologic Studies Depression Scale (CES-D), is a 20-item measure that asks respondents to rate how often over the past week they experienced symptoms associated with depression on a scale from 0 to 3 (0 = "Rarely or None of the Time," 1 = "Some or Little of the Time," 2 = "Moderately or Much of the time," 3 = "Most or Almost All the Time"). Scores are summed and range from 0 to 60, with high scores indicating greater depressive symptoms.
Depressive symptoms: Changes in depressive symptoms | Baseline to 6-months post-intervention
  Center for Epidemiologic Studies Depression Scale (CES-D), is a 20-item measure that asks respondents to rate how often over the past week they experienced symptoms associated with depression on a scale from 0 to 3 (0 = "Rarely or None of the Time," 1 = "Some or Little of the Time," 2 = "Moderately or Much of the time," 3 = "Most or Almost All the Time"). Scores are summed and range from 0 to 60, with high scores indicating greater depressive symptoms.
Depressive symptoms: Changes in depressive symptoms | Baseline to 12-months post-intervention
  Center for Epidemiologic Studies Depression Scale (CES-D), is a 20-item measure that asks respondents to rate how often over the past week they experienced symptoms associated with depression on a scale from 0 to 3 (0 = "Rarely or None of the Time," 1 = "Some or Little of the Time," 2 = "Moderately or Much of the time," 3 = "Most or Almost All the Time"). Scores are summed and range from 0 to 60, with high scores indicating greater depressive symptoms.
Generalized Anxiety: Changes in symptoms of generalized anxiety | Baseline to Day 7 post-transplant
  Generalized Anxiety Disorder Screener (GAD-7), which measures generalized anxiety symptoms in the past 7 days with 7 items rated on a 0-3 scale (0="Not at all," 1="Several days," 2="More than half the days," 3="Nearly every day"). Scores are summed and range from 0 to 21, with higher scores indicating greater symptomatology.
Generalized Anxiety: Changes in symptoms of generalized anxiety | Baseline to Day 14 post-transplant
  Generalized Anxiety Disorder Screener (GAD-7), which measures generalized anxiety symptoms in the past 7 days with 7 items rated on a 0-3 scale (0="Not at all," 1="Several days," 2="More than half the days," 3="Nearly every day"). Scores are summed and range from 0 to 21, with higher scores indicating greater symptomatology.
Generalized Anxiety: Changes in symptoms of generalized anxiety | Baseline to 1-week post-intervention
  Generalized Anxiety Disorder Screener (GAD-7), which measures generalized anxiety symptoms in the past 7 days with 7 items rated on a 0-3 scale (0="Not at all," 1="Several days," 2="More than half the days," 3="Nearly every day"). Scores are summed and range from 0 to 21, with higher scores indicating greater symptomatology.
Generalized Anxiety: Changes in symptoms of generalized anxiety | Baseline to 3-months post-intervention
  Generalized Anxiety Disorder Screener (GAD-7), which measures generalized anxiety symptoms in the past 7 days with 7 items rated on a 0-3 scale (0="Not at all," 1="Several days," 2="More than half the days," 3="Nearly every day"). Scores are summed and range from 0 to 21, with higher scores indicating greater symptomatology.
Generalized Anxiety: Changes in symptoms of generalized anxiety | Baseline to 6-months post-intervention
  Generalized Anxiety Disorder Screener (GAD-7), which measures generalized anxiety symptoms in the past 7 days with 7 items rated on a 0-3 scale (0="Not at all," 1="Several days," 2="More than half the days," 3="Nearly every day"). Scores are summed and range from 0 to 21, with higher scores indicating greater symptomatology.
Generalized Anxiety: Changes in symptoms of generalized anxiety | Baseline to 12-months post-intervention
  Generalized Anxiety Disorder Screener (GAD-7), which measures generalized anxiety symptoms in the past 7 days with 7 items rated on a 0-3 scale (0="Not at all," 1="Several days," 2="More than half the days," 3="Nearly every day"). Scores are summed and range from 0 to 21, with higher scores indicating greater symptomatology.
Cancer-specific anxiety: Changes in symptoms of cancer-specific anxiety | Baseline to Day 7 post-transplant
  Impact of event scale (IES), which includes 15 items that assess difficulties (intrusive thoughts and feelings, avoidance) caused by a traumatic event (in this study, the diagnosis and transplant). Respondents rate how much they were distressed or bothered by each difficulty during the past 7 days using a 5-point scale ranging from 0 ("not at all") to 4 ("extremely"). Responses are summed to give a total score ranging from 0 to 60, with higher scores indicating greater symptomatology.
Cancer-specific anxiety: Changes in symptoms of cancer-specific anxiety | Baseline to Day 14 post-transplant
  Impact of event scale (IES), which includes 15 items that assess difficulties (intrusive thoughts and feelings, avoidance) caused by a traumatic event (in this study, the diagnosis and transplant). Respondents rate how much they were distressed or bothered by each difficulty during the past 7 days using a 5-point scale ranging from 0 ("not at all") to 4 ("extremely"). Responses are summed to give a total score ranging from 0 to 60, with higher scores indicating greater symptomatology.
Cancer-specific anxiety: Changes in symptoms of cancer-specific anxiety | Baseline to 1-week post-intervention
  Impact of event scale (IES), which includes 15 items that assess difficulties (intrusive thoughts and feelings, avoidance) caused by a traumatic event (in this study, the diagnosis and transplant). Respondents rate how much they were distressed or bothered by each difficulty during the past 7 days using a 5-point scale ranging from 0 ("not at all") to 4 ("extremely"). Responses are summed to give a total score ranging from 0 to 60, with higher scores indicating greater symptomatology.
Cancer-specific anxiety: Changes in symptoms of cancer-specific anxiety | Baseline to 3-months post-intervention
  Impact of event scale (IES), which includes 15 items that assess difficulties (intrusive thoughts and feelings, avoidance) caused by a traumatic event (in this study, the diagnosis and transplant). Respondents rate how much they were distressed or bothered by each difficulty during the past 7 days using a 5-point scale ranging from 0 ("not at all") to 4 ("extremely"). Responses are summed to give a total score ranging from 0 to 60, with higher scores indicating greater symptomatology.
Cancer-specific anxiety: Changes in symptoms of cancer-specific anxiety | Baseline to 6-months post-intervention
  Impact of event scale (IES), which includes 15 items that assess difficulties (intrusive thoughts and feelings, avoidance) caused by a traumatic event (in this study, the diagnosis and transplant). Respondents rate how much they were distressed or bothered by each difficulty during the past 7 days using a 5-point scale ranging from 0 ("not at all") to 4 ("extremely"). Responses are summed to give a total score ranging from 0 to 60, with higher scores indicating greater symptomatology.
Cancer-specific anxiety: Changes in symptoms of cancer-specific anxiety | Baseline to 12-months post-intervention
  Impact of event scale (IES), which includes 15 items that assess difficulties (intrusive thoughts and feelings, avoidance) caused by a traumatic event (in this study, the diagnosis and transplant). Respondents rate how much they were distressed or bothered by each difficulty during the past 7 days using a 5-point scale ranging from 0 ("not at all") to 4 ("extremely"). Responses are summed to give a total score ranging from 0 to 60, with higher scores indicating greater symptomatology.
Quality of life: Changes in quality of life | Baseline to Day 7 post-transplant
  Patient-reported Outcomes Measurement Information System (PROMIS) V1.2 Global Health measure, which includes 10 items assessing the domains of physical and mental health functioning, rated on a scale from 1-5 or 0 to 10, with specific responses differing across items. Items are summed and conversion tables are used to convert the simple summed raw scores into T-score values for each respondent. T-Score distributions are standardized such that a 50 represents the average (mean) for the US general population, and the standard deviation around that mean is 10 points. Higher scores indicate better quality of life
Quality of life: Changes in quality of life | Baseline to Day 14 post-transplant
  Patient-reported Outcomes Measurement Information System (PROMIS) V1.2 Global Health measure, which includes 10 items assessing the domains of physical and mental health functioning, rated on a scale from 1-5 or 0 to 10, with specific responses differing across items. Items are summed and conversion tables are used to convert the simple summed raw scores into T-score values for each respondent. T-Score distributions are standardized such that a 50 represents the average (mean) for the US general population, and the standard deviation around that mean is 10 points. Higher scores indicate better quality of life
Quality of life: Changes in quality of life | Baseline to 1-week post-intervention
  Patient-reported Outcomes Measurement Information System (PROMIS) V1.2 Global Health measure, which includes 10 items assessing the domains of physical and mental health functioning, rated on a scale from 1-5 or 0 to 10, with specific responses differing across items. Items are summed and conversion tables are used to convert the simple summed raw scores into T-score values for each respondent. T-Score distributions are standardized such that a 50 represents the average (mean) for the US general population, and the standard deviation around that mean is 10 points. Higher scores indicate better quality of life
Quality of life: Changes in quality of life | Baseline to 3-months post-intervention
  Patient-reported Outcomes Measurement Information System (PROMIS) V1.2 Global Health measure, which includes 10 items assessing the domains of physical and mental health functioning, rated on a scale from 1-5 or 0 to 10, with specific responses differing across items. Items are summed and conversion tables are used to convert the simple summed raw scores into T-score values for each respondent. T-Score distributions are standardized such that a 50 represents the average (mean) for the US general population, and the standard deviation around that mean is 10 points. Higher scores indicate better quality of life
Quality of life: Changes in quality of life | Baseline to 6-months post-intervention
  Patient-reported Outcomes Measurement Information System (PROMIS) V1.2 Global Health measure, which includes 10 items assessing the domains of physical and mental health functioning, rated on a scale from 1-5 or 0 to 10, with specific responses differing across items. Items are summed and conversion tables are used to convert the simple summed raw scores into T-score values for each respondent. T-Score distributions are standardized such that a 50 represents the average (mean) for the US general population, and the standard deviation around that mean is 10 points. Higher scores indicate better quality of life
Quality of life: Changes in quality of life | Baseline to 12-months post-intervention
  Patient-reported Outcomes Measurement Information System (PROMIS) V1.2 Global Health measure, which includes 10 items assessing the domains of physical and mental health functioning, rated on a scale from 1-5 or 0 to 10, with specific responses differing across items. Items are summed and conversion tables are used to convert the simple summed raw scores into T-score values for each respondent. T-Score distributions are standardized such that a 50 represents the average (mean) for the US general population, and the standard deviation around that mean is 10 points. Higher scores indicate better quality of life
Fatigue: Changes in fatigue | Baseline to Day 7 post-transplant
  Functional Assessment of Chronic Illness Therapy-Fatigue (FACIT-Fatigue), which measures level of fatigue in the past 7 days with 13 items rated on a 0-4 scale (0="Not at all," 1="A little bit," 2="Somewhat," 3="Quite a bit," 4="Very much"). Eleven responses are reverse scored and responses are then averaged to yield a scale ranging from 0 to 52, in which higher scores indicate lower fatigue.
Fatigue: Changes in fatigue | Baseline to Day 14 post-transplant
  Functional Assessment of Chronic Illness Therapy-Fatigue (FACIT-Fatigue), which measures level of fatigue in the past 7 days with 13 items rated on a 0-4 scale (0="Not at all," 1="A little bit," 2="Somewhat," 3="Quite a bit," 4="Very much"). Eleven responses are reverse scored and responses are then averaged to yield a scale ranging from 0 to 52, in which higher scores indicate lower fatigue.
Fatigue: Changes in fatigue | Baseline to 1-week post-intervention
  Functional Assessment of Chronic Illness Therapy-Fatigue (FACIT-Fatigue), which measures level of fatigue in the past 7 days with 13 items rated on a 0-4 scale (0="Not at all," 1="A little bit," 2="Somewhat," 3="Quite a bit," 4="Very much"). Eleven responses are reverse scored and responses are then averaged to yield a scale ranging from 0 to 52, in which higher scores indicate lower fatigue.
Fatigue: Changes in fatigue | Baseline to 3-month post-intervention
  Functional Assessment of Chronic Illness Therapy-Fatigue (FACIT-Fatigue), which measures level of fatigue in the past 7 days with 13 items rated on a 0-4 scale (0="Not at all," 1="A little bit," 2="Somewhat," 3="Quite a bit," 4="Very much"). Eleven responses are reverse scored and responses are then averaged to yield a scale ranging from 0 to 52, in which higher scores indicate lower fatigue.
Fatigue: Changes in fatigue | Baseline to 6-month post-intervention
  Functional Assessment of Chronic Illness Therapy-Fatigue (FACIT-Fatigue), which measures level of fatigue in the past 7 days with 13 items rated on a 0-4 scale (0="Not at all," 1="A little bit," 2="Somewhat," 3="Quite a bit," 4="Very much"). Eleven responses are reverse scored and responses are then averaged to yield a scale ranging from 0 to 52, in which higher scores indicate lower fatigue.
Fatigue: Changes in fatigue | Baseline to 12-month post-intervention
  Functional Assessment of Chronic Illness Therapy-Fatigue (FACIT-Fatigue), which measures level of fatigue in the past 7 days with 13 items rated on a 0-4 scale (0="Not at all," 1="A little bit," 2="Somewhat," 3="Quite a bit," 4="Very much"). Eleven responses are reverse scored and responses are then averaged to yield a scale ranging from 0 to 52, in which higher scores indicate lower fatigue.

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Lombardi Comprehensive Cancer Center at Georgetown University Medical Center, Washington D.C., District of Columbia
  - Robert H. Lurie Comprehensive Cancer Center at Northwestern University, Chicago, Illinois
  - John Theurer Cancer Center at Hackensack University Medical Center, Hackensack, New Jersey

IPD SHARING:
Plan to Share IPD: No
All IPD will be protected and maintained by the study team

REFERENCES:
- [Derived] Whitmore L, Schulte T, Bovbjerg K, Hartstein M, Austin J, Luta G, McFarland L, Rowley SD, Nyirenda T, Lewis-Thames M, Stanton AL, Valdimarsdottir H, Graves K, Rini C. Efficacy of expressive helping in adult hematologic cancer patients undergoing stem cell transplant: protocol for the Writing for Insight, Strength, and Ease (WISE) study's two-arm randomized controlled trial. Trials. 2021 Oct 20;22(1):722. doi: 10.1186/s13063-021-05676-w. PMID 34670600

DOCUMENTS (1):
  • Informed Consent Form (2021-08-23): https://cdn.clinicaltrials.gov/large-docs/58/NCT03800758/ICF_000.pdf